CLINICAL TRIAL: NCT05844176
Title: Intracranial Arterial Stenosis in Young Patients: a Multicenter Longitudinal Cohort Study
Brief Title: Intracranial Arterial Stenosis in Young Patients
Acronym: ICAS-Young
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Other Study IDs: ICAS-Young
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Intracranial Arterial Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic intracranial arterial stenosis
  Interventions: Other: Routine clinical treatment
- Asymptomatic intracranial arterial stenosis
  Interventions: Other: Routine clinical treatment

INTERVENTIONS:
Other: Routine clinical treatment — Routine clinical treatment is based on the latest international and local guidelines

SUMMARY:
The goal of this study is to evaluate the characteristic of intracranial arterial stenosis among young patients.

ELIGIBILITY:
Inclusion Criteria:

* age < 45 years.
* stenosis of a major intracranial artery.

Exclusion Criteria:

-

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with intracranial arterial stenosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke in territory of qualifying artery | 1 year

SECONDARY OUTCOMES:
Ischemic stroke in other territory | 1 year
Any stroke | 1 year
Death | 1 year
Stenosis of the intracranial artery | 1 year

OTHER OUTCOMES:
Ischemic stroke in the territory of qualifying artery | 3 year
Ischemic stroke in other territory | 3 year
Any stroke | 3 year
Death | 3 year
Stenosis of the intracranial artery | 3 year
Ischemic stroke in the territory of qualifying artery | 5 year
Ischemic stroke in other territory | 5 year
Any stroke | 5 year
Death | 5 year
Stenosis of the intracranial artery | 5 year

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Suzhou Municipal Hoapital, Suzhou, Anhui
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xuanwu Hospital, Capital Medical University, Beijing
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou